CLINICAL TRIAL: NCT03895567
Title: A Randomised Crossover Study of the Pharmacokinetics, Safety and Tolerability of Two Rectal Formulations of Ceftriaxone Compared to Parenteral Ceftriaxone, in Healthy Thai Adults.
Brief Title: Study to Compare Blood Levels of Ceftriaxone Given by Suppository or Injection.
Acronym: CefREC
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was suspended while the researchers secured new funding.
Sponsor: University of Oxford (Other)
Collaborators: Biopharma (Orofino Pharmaceuticals Group) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BAC18003
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- ABC (Experimental): A. Ceftriaxone (Roche ®) 500mg (slow intravenous injection) B. Ceftriaxone rectal dosage form test formulation 1- hard-shell gelatin capsule (1 x 500mg) C. Ceftriaxone rectal dosage form test formulation 2- rectodispersible mannitol-based tablet (1 x 500mg)
  Interventions: Drug: A. Ceftriaxone (Roche ®) 500mg (slow intravenous injection); Drug: B. Ceftriaxone rectal dosage form test formulation 1 (1 x 500mg); Drug: C. Ceftriaxone rectal dosage form test formulation 2 (1 x 500mg)
- ACB (Experimental): A. Ceftriaxone (Roche ®) 500mg (slow intravenous injection) C. Ceftriaxone rectal dosage form test formulation 2- rectodispersible mannitol-based tablet (1 x 500mg) B. Ceftriaxone rectal dosage form test formulation 1- hard-shell gelatin capsule (1 x 500mg)
  Interventions: Drug: A. Ceftriaxone (Roche ®) 500mg (slow intravenous injection); Drug: B. Ceftriaxone rectal dosage form test formulation 1 (1 x 500mg); Drug: C. Ceftriaxone rectal dosage form test formulation 2 (1 x 500mg)
- BAC (Experimental): B. Ceftriaxone rectal dosage form test formulation 1- hard-shell gelatin capsule (1 x 500mg) A. Ceftriaxone (Roche ®) 500mg (slow intravenous injection) C. Ceftriaxone rectal dosage form test formulation 2- rectodispersible mannitol-based tablet (1 x 500mg)
  Interventions: Drug: A. Ceftriaxone (Roche ®) 500mg (slow intravenous injection); Drug: B. Ceftriaxone rectal dosage form test formulation 1 (1 x 500mg); Drug: C. Ceftriaxone rectal dosage form test formulation 2 (1 x 500mg)
- BCA (Experimental): B. Ceftriaxone rectal dosage form test formulation 1- hard-shell gelatin capsule (1 x 500mg) C. Ceftriaxone rectal dosage form test formulation 2- rectodispersible mannitol-based tablet (1 x 500mg) A. Ceftriaxone (Roche ®) 500mg (slow intravenous injection)
  Interventions: Drug: A. Ceftriaxone (Roche ®) 500mg (slow intravenous injection); Drug: B. Ceftriaxone rectal dosage form test formulation 1 (1 x 500mg); Drug: C. Ceftriaxone rectal dosage form test formulation 2 (1 x 500mg)
- CAB (Experimental): C. Ceftriaxone rectal dosage form test formulation 2- rectodispersible mannitol-based tablet (1 x 500mg) A. Ceftriaxone (Roche ®) 500mg (slow intravenous injection) B. Ceftriaxone rectal dosage form test formulation 1- hard-shell gelatin capsule (1 x 500mg)
  Interventions: Drug: A. Ceftriaxone (Roche ®) 500mg (slow intravenous injection); Drug: B. Ceftriaxone rectal dosage form test formulation 1 (1 x 500mg); Drug: C. Ceftriaxone rectal dosage form test formulation 2 (1 x 500mg)
- CBA (Experimental): C. Ceftriaxone rectal dosage form test formulation 2- rectodispersible mannitol-based tablet (1 x 500mg) B. Ceftriaxone rectal dosage form test formulation 1- hard-shell gelatin capsule (1 x 500mg) A. Ceftriaxone (Roche ®) 500mg (slow intravenous injection)
  Interventions: Drug: A. Ceftriaxone (Roche ®) 500mg (slow intravenous injection); Drug: B. Ceftriaxone rectal dosage form test formulation 1 (1 x 500mg); Drug: C. Ceftriaxone rectal dosage form test formulation 2 (1 x 500mg)

INTERVENTIONS:
Drug: A. Ceftriaxone (Roche ®) 500mg (slow intravenous injection) — Parenteral ceftriaxone
  Intravenous injection of 500mg of ceftriaxone sodium (Rocephin®; Roche).
Drug: B. Ceftriaxone rectal dosage form test formulation 1 (1 x 500mg) — Rectal ceftriaxone formulations
  Formulation 1 ceftriaxone 500mg + Na-CDC 125mg hard-shell gelatin capsule
Drug: C. Ceftriaxone rectal dosage form test formulation 2 (1 x 500mg) — Rectal ceftriaxone formulations
  Formulation 2 ceftriaxone 500mg + Na-CDC 125mg rectodispersible mannitol-based tablet

SUMMARY:
Phase 1, three-way cross-over, randomised, open label comparison of intravenous versus two rectal dosage forms of ceftriaxone in 37 healthy Thai adults.

The following regimens will be evaluated in random order in all participants:

A. Ceftriaxone (Roche ®) 500mg (slow intravenous injection) B. Ceftriaxone rectal dosage form test formulation 1-hard-shell gelatin capsule (1 x 500mg) C. Ceftriaxone rectal dosage form test formulation 2-rectodispersible mannitol-based tablet (1 x 500mg)

Possible schedules: ABC, ACB, BAC, BCA, CAB, CBA. Each recipient will receive a single treatment dose of each of the three formulations in an order predetermined by a computer generated randomisation list. This will be a constrained randomization which ensures approximately balanced proportions for all six schedules (either 6 or 7 participants per schedule). There will be 7-28 days washout period between doses. The last follow up visit is 28 (+ 2) days after final dose. Participants lost to follow-up or unevaluable for any reason before completion of pharmacokinetic sampling after the final dose will be replaced at the discretion of the investigators with another participant of the same population, if either sample size or completeness of dataset is compromised.

This study is funded by the Medical Research Council. The grant reference number is MR/W021560/1

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female, aged 18 to 46 years (inclusive)
* Willing and able to give informed consent to participate in the trial
* Able, in the investigators opinion, and willing to comply with the study requirements and followup.

Exclusion Criteria:

* Female participant who is pregnant, lactating or planning pregnancy during the course of the study.
* Presence of any condition which in the judgment of the investigator would affect the absorption of the rectal formulation e.g. previous surgery, haemorrhoids, inflammatory bowel disease
* Irritable bowel syndrome (IBS) or diarrhoea in the 24 hours prior to study drug administration
* Presence of any condition which in the judgment of the investigator would place the participant at undue risk or interfere with the results of the study (e.g. serious underlying cardiac, renal, hepatic or neurological disease; severe malnutrition; congenital defects or febrile condition).
* Seropositive for HIV at screening
* Hepatitis B surface antigen (HBsAg) detected in serum at screening.
* Seropositive for hepatitis C virus (antibodies to HCV) at screening
* Participation in a clinical trial and/or has received a drug or a new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of study medication and throughout the study period.
* Any medical condition that in the judgment of the investigator would make the administration of the study treatments unsafe.
* Use of medications known to have a potentially clinically significant interaction with ceftriaxone or with sodium chenodeoxycholate (Na-CDC) in the 28 days prior to the first dose and throughout the study period. This includes aluminium-containing antacids, colestipol, phenobarbital and the combined oral contraceptive pill.
* Known 27-hydroxylase deficiency (presenting as cerebrotendinous xanthomatosis)
* History of anaphylaxis and /or hypotension, laryngeal oedema, wheezing, angioedema or urticarial rash following treatment with ceftriaxone, another cephalosporin or any beta lactam (e.g. penicillin).
* History of any other clinically significant reaction to ceftriaxone, another cephalosporin or beta lactam e.g. drug induced nephritis, hepatitis, erythema multiforme that, in the opinion of the investigator, contraindicates participation in the study.
* Serious chronic illness.
* Abnormal baseline laboratory screening test as defined below:

  * AST > 2 x upper normal limit
  * ALT > 2 x upper normal limit
  * Anaemia (Hb < 11 g/dL for female and Hb < 12 g/dL for male),
  * Platelets < 150,000
  * Total bilirubin > 2 x upper normal limit
* Hepatomegaly, right upper quadrant abdominal pain or tenderness.
* Body Mass Index> 35
* History of alcohol or substance abuse or dependence during the 6 months before study participation: History of regular alcohol consumption averaging >7 drinks/week for women or >14 drinks/week for men. One drink is equivalent to 12 g alcohol = 5 oz (150 mL) of wine or 12 oz (360 mL) of beer or 1.5 oz (45 mL) of 80 proof distilled spirits.

Ages: 18 Years to 46 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Estimated)
Dates: Start 2026-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Bioavailablity of rectal formulation | Approximately 9 months

SECONDARY OUTCOMES:
Description of Exposure (AUC0-∞) | Approximately 9 months
Description of Peak concentration (Cmax) | Approximately 100 days
Description of Absorption rate (Tmax) | Approximately 9 months
Time above a plasma concentration of 1µg/mL (this concentration is above the MIC90 for major neonatal pathogens and is the lower limit of detection of the assay) | Approximately 9 months
Occurrence of serious adverse events (SAEs) from the date of the first dose to 28 days after the final dose, according to the MedDRA classification. | Approximately 9 months
Occurrence of all adverse events from the date of the first dose to 28 days after the final dose, according to the MedDRA classification. | Approximately 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Ashley, MD, Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (1):
- Faculty of Tropical Medicine, Mahidol University, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
With participant's consent, participant's clinical data and results from blood analyses stored in our database may be shared with Biopharma Orofino Pharmaceuticals Group, regulatory authorities, or other researchers to use in the future. However, the other researchers will not be given any information that could identify the participant.
Supporting Information: Study Protocol
Access Criteria: Requests to share data will be considered by the MORU data access committee in line with the MORU data sharing policy
URL: https://www.tropmedres.ac/units/moru-bangkok/bioethics-engagement/data-sharing